CLINICAL TRIAL: NCT00309348
Title: New Doppler Instrument for Preventing Impending Access-Graft Failure Randomized Trial
Brief Title: Ultrasound Instrument to Prevent Dialysis Graft Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DVX, LLC (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44DK067775 (NIH); R44DK067775 (NIH)
Record Dates: First submitted 2006-03-30; First posted 2006-03-31 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly measurement of graft flow (Experimental): The surveillance group was measured with the FloMon instrument weekly, and all procedures related to their access-grafts recorded
  Interventions: Other: Weekly measurement of graft flow
- Control (No Intervention): The control group was questioned weekly with regard to their graft status and whether there had been any graft-related procedures

INTERVENTIONS:
Other: Weekly measurement of graft flow
  Arms: Weekly measurement of graft flow

SUMMARY:
This research study aims to show that a newly developed investigational Doppler instrument can reliably measure blood flow in dialysis access grafts, to see if a decrease in the flow may be a sign of impending graft failure and also to see if there is evidence that by monitoring the flow in these grafts their lives may be extended.

The new investigational device is to be known as FloMon; this is an ultrasonic device that provides blood flow measurements from a small probe placed in a noninvasive manner above the graft or blood vessel. The instrument is being developed so that it may help give insight to on-coming graft failure which may be prevented.

The FloMon is an extension of a previously Food and Drug Administration (FDA) cleared instrument, Echoflow-A, which had been used in a similar study as this one. The Echoflow-A is similar to this device in all respects with the exception of design and calculation of measurement. The FloMon compared to the Echoflow-A is better ergonomically designed and reads flow readings in about 2 minutes versus twice the time necessary to take similar measurements using the Echoflow-A.

DETAILED DESCRIPTION:
Vascular access failure is one of the largest causes of morbidity for chronic hemodialysis patients: 16-25% of hospital admissions among United States end-stage renal disease (ESRD) patients are related to vascular access complications, and the associated cost is estimated to be over one billion dollars per year.

The most frequent cause of AV access-graft failure is thrombosis that occurs as a result of stenosis at or near the venous anastomosis. Over 50% of existing vascular access-grafts in the US are 6 mm PTFE tubes and their thrombosis rate is much higher than that of native Arteriovenous Fistulas (AVF).

Several studies have shown that early detection and repair of stenosis can prevent access thrombosis, reducing the morbidity and costs that follow thrombosis. The cost of duplex ultrasound for access monitoring is prohibitive. Blood flow, measured by indicator-dilution methods, seems to be a reliable indicator of impending access failure, but recent randomized controlled studies intended to examine this were equivocal.

This study, funded by the NIH (2R44 DK067775), is to determine if a new instrument to monitor access blood-flow can reduce graft failure and associated costs. In a pilot study using the new Doppler ultrasound instrument for weekly monitoring, conducted by the Renal Research Institute and funded by the NIH, the method predicted impending graft failure with 80% sensitivity and a false-alarm rate of less than .5/year. It measures access blood flow in less than three minutes, and uses almost no consumables.

This study is designed to test if monitoring with the new instrument improves health and reduces cost for hemodialysis patients with access-grafts.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients with an AV access graft

Exclusion Criteria:

* Anticipated change in renal replacement modality or geographic location
* Inability to give informed consent
* Anticipated life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-02-27 (Actual); Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

PRIMARY OUTCOMES:
Number of low flow events | Mean follow-up of 15 months
  A "Low-Flow Event" is an intervention, whether an angioplasty or thrombectomy, to increase graft flow.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Levine, MD, Principal Investigator — Renal Research Institute; David Vilkomerson, PhD, Principal Investigator — DVX, LLC
Locations (2):
- United States (2):
  - Queens Artificial Kidney Center, Jackson Heights, New York
  - St Albans Dialysis Center, Jamaica, New York